CLINICAL TRIAL: NCT02927340
Title: A Phase II Study of Lorlatinib (PF-06463922) in Advanced Anaplastic Lymphoma Kinase (ALK) and ROS Proto-Oncogene 1 (ROS1) Rearranged Non-Small Cell Lung Cancer (NSCLC) With Central Nervous System (CNS) Metastasis in the Absence of Measurable Extracranial Lesions
Brief Title: A Study of Lorlatinib in Advanced ALK and ROS1 Rearranged Lung Cancer With CNS Metastasis in the Absence of Measurable Extracranial Lesions
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ibiayi Dagogo-Jack, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-248
Record Dates: First submitted 2016-09-26; First posted 2016-10-07 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-01

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — lorlatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lorlatinib (Experimental): Lorlatinib will be administered orally once daily on a 21 day cycle Blood will be collected for biomarker studies
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib

SUMMARY:
This research study is studying a drug as a possible treatment for ALK-positive or ROS1-positive non-small cell lung cancer (NSCLC).

The following drug will be involved in this study :

* Lorlatinib

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied. The FDA (the U.S. Food and Drug Administration) has not approved Lorlatinib as a treatment for any disease.

All participants in this study will receive Lorlatinib. Lorlatinib targets the abnormal ALK or ROS1 proteins in NSCLC cells. Lorlatinib has been tested in other research studies and results show that the medicine may help to control the growth of NSCLC even after it has spread to the CNS. The CNS is a term used to refer to the brain and spinal cord, including the lining of the brain and spinal cord which is called the meninges.

In this research study, the investigators are trying to determine whether lorlatinib is effective in controlling the growth of cancer cells after they have spread to the CNS. Another purpose of this study is to determine why the cancer cells that have spread to the participant CNS have continued to grow despite treatment with other drugs. For this reason, blood samples will be collected as part of this study to assess the DNA released by the participants cancer cells into their blood when the cells travel to other sites in their body.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of metastatic NSCLC (Stage IV, American Joint Committee on Cancer v7.0) that carries an ALK rearrangement, as determined by the Food and Drug Administration (FDA)-approved FISH test, using Vysis® ALK Break apart fluorescence in situ hybridization (FISH) Probe Kit (defined as 15% or more positive tumor cells), or the Ventana® immunohistochemistry (IHC) test, or a ROS1 rearrangement as determined by FISH or reverse transcription polymerase chain reaction (RT-PCR) or Next Generation Sequencing (NGS) via a local diagnostic test (LDT).
* ALK positive NSCLC patients must either be treatment naive in the advanced setting or have had disease progression on or intolerance to at least 1 previous ALK inhibitor. ROS1 positive NSCLC patients must either be treatment naive in the advanced setting or have had disease progression on or intolerance to at least 1 previous ROS1 inhibitor.
* Presence of radiographically suspected leptomeningeal disease (LM) or carcinomatous meningitis (CM) AND/OR presence of at least one CNS lesion for which the following criteria are met:

  * For patients without leptomeningeal disease: presence of at least one parenchymal CNS lesion that is at least 5 mm in size. Note: Intra-cranial disease assessments can only be performed using contrast-enhanced magnetic resonance imaging (MRI). MRI scan slices of 1 mm are necessary for brain metastases between 5 and 10 mm in size.
  * The lesion(s) must be newly diagnosed or be present as progression after local therapy, including surgery and/or radiation therapy. For patients who have received local therapy, progression of pre-existing lesions based on RECIST v1.1 (>20% increase in longest diameter on baseline scan) or new lesions are required.
  * Participants who are receiving corticosteroids must be on a stable or decreasing dose for at least 2 weeks prior to the first dose of study treatment.
  * For patients with suspected LM or CM based on imaging, spinal fluid sampling for confirmation is not required. For patients who do undergo spinal fluid sampling, those with negative spinal fluid (CSF) are eligible to enter.
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥60%)
* Life expectancy of ≥ 12 weeks, in the opinion of the investigator
* Adequate hematologic function, including:

  * Platelet count ≥ 100 x 109/L
  * Absolute neutrophil count (ANC) ≥ 1,500/µL
  * Hemoglobin ≥ 9 g/dL
* Adequate renal function, including:

  * Serum creatinine ≤1.5x the upper limit of normal (ULN) or an estimated glomerular filtration rate (eGFR) calculated using the Modification of Diet in Renal Disease (MDRD) equation of at least 45 mL/min/1.73 m2
* Adequate pancreatic function, including:

  * Serum lipase ≤ 1.5x ULN
* Adequate liver function, including:

  * Total serum bilirubin ≤ 1.5x ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0x ULN in the absence of known metastatic involvement of the liver or AST and ALT ≤ 5.0x ULN if there is metastatic liver involvement.
  * Alkaline phosphatase ≤ 2.5x ULN in the absence of known bone metastases or ≤ 5.0x ULN in the case of bone metastases.
* After progression on or intolerance to prior ALK or ROS inhibitor therapy:

  * A minimum washout period of at least 5 half-lives between the last dose of ALK or ROS inhibitor therapy and the first dose of study treatment is required. A shorter washout period may be considered in the event of disease flare, after discussion with the Sponsor.
  * Patients must have recovered from treatment toxicities to ≤ Grade 1 or to their pretreatment levels except for adverse events (AEs) that in the investigator's judgment do not constitute a safety risk for the patient.
* Patients can either be chemotherapy-naive or have received at least one line of platinum-based chemotherapy for locally advanced or metastatic disease. Acute effects of therapy must have resolved to baseline severity or to CTCAE grade ≤1 except for AEs that in the investigator's judgment do not constitute a safety risk for the patient.
* Recovery from effects of any major surgery or significant traumatic injury at least 28 days before the first dose of study treatment
* For all women of childbearing potential, a negative pregnancy test must be obtained at the baseline visit before starting study treatment.

  * For women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use two adequate methods of contraception, including at least one method with a failure rate of < 1% per year, during the treatment period and for at least 90 days after the last dose of study drug.
  * Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  * Examples of contraceptive methods with a failure rate of < 1% per year include tubal ligation, male sterilization, hormonal implants, established, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices. Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of <1% per year. Barrier methods must always be supplemented with the use of a spermicide.
  * For men: agreement to remain abstinent or use a barrier method of contraception (e.g., condom) during the treatment period and for at least 90 days after the last dose of study drug and agreement to refrain from donating sperm during this same period
  * Men with a pregnant partner must agree to remain abstinent or use a condom for the duration of the pregnancy.
  * Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior use of lorlatinib (PF-06463922)
* Presence of measurable extracranial disease by RECIST v1.1
* Spinal cord compression is excluded unless the patient demonstrates good pain control attained through therapy and there is stabilization or recovery of neurological function for two weeks prior to study entry.
* Major surgery within 4 weeks of study entry. Minor surgical procedures (eg port insertion, pleurex catheter placement) are not excluded, but sufficient time should have passed for wound healing.
* Radiation therapy (except palliative to relieve bone pain) within 7 days of study entry. Palliative radiation (≤ 10 fractions) must have been completed at least 48 hours prior to study entry. Stereotactic or small field brain irradiation must have been completed at least 7 days prior to study entry. Whole brain radiation must have been completed at least 2 weeks prior to study entry.
* Systemic anti-cancer therapy completed within a minimum of 5 half-lives of study entry.
* Active and clinically significant bacterial, fungal, or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
* Any one of the following currently or in the previous 3 months: myocardial infarction, congenital long QT syndrome, Torsades de Pointes, uncontrolled arrhythmias (including sustained ventricular tachyarrhythmia and ventricular fibrillation), right bundle branch block and left anterior fascicular hemiblock (bifascicular block), unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (CHF New York Heart Association Classification III or IV) , cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism not adequate medically managed with anticoagulants, ongoing cardiac dysrhythmias of CTCAE grade ≥ 2, symptomatic atrial fibrillation of any grade, corrected QT (QTc) interval ≥ 481 msec at screening
* Patients with predisposing characteristics for acute pancreatitis according to investigator judgment (eg current gallstone disease, alcoholism)
* History of extensive, disseminated, bilateral or presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease including pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis and pulmonary fibrosis. Patients with history of prior radiation pneumonitis are not excluded.
* Participants who are receiving any other investigational agents.
* Active inflammatory gastrointestinal disease or previous gastric resection or lap band.
* Pregnant or lactating women
* Patients with a history of organ transplant including high dose chemotherapy with autologous stem cell rescue
* Current use or anticipated need for food or drugs that are known strong or moderate CYP3A4 inhibitors, including their administration within 10 days prior to the first lorlatinib dose (ie, strong CYP3A4 inhibitors: grapefruit juice or grapefruit/grapefruit related citrus fruits [eg, Seville oranges, pomelos], ketoconazole, miconazole, itraconazole, voriconazole, posaconazole, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, amprenavir, fosamprenavir nefazodone, lopinavir, troleandomycin, mibefradil, and conivaptan; Moderate CYP3A4 inhibitors: erythromycin, verapamil, atazanavir, delavirdine, fluconazole, darunavir, diltiazem, aprepitant, imatinib, tofisopam, ciprofloxacin, cimetidine)
* Current use or anticipated need for drugs that are known strong CYP3A4 inducers, including their administration within 12 days prior to the first lorlatinib dose (ie, phenobarbital, rifampin, phenytoin, carbamazepine, rifabutin, rifapentin, clevidipine, St. John's Wort).
* Concurrent use of drugs that are CYP3A4 substrates with narrow therapeutic indices such as astemizole, terfenadine, cisapride, pimozide, quinidine, tacrolimus, cyclosporine, sirolimus, (alfentanil and fentanyl, including transdermal patch) or ergot alkaloids (ergotamine, dihydroergotamine) is not permitted or caution is warranted.
* Concurrent use of drugs that are CYP2C9 substrates with narrow therapeutic indices, such as warfarin, phenytoin or a sensitive substrate such as celecoxib is not permitted or caution is warranted.
* Concurrent use of drugs that are sensitive CYP2B6 substrates, such as bupropion, efavirenz is not permitted or caution is warranted.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lorlatinib.

Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2022-01 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Intracranial Disease Control Rate (DCR) | 12 weeks
  DCR will be calculated at 12 weeks based on response assessments in the brain for patients with measurable CNS disease

SECONDARY OUTCOMES:
Median intracranial Progression-Free Survival (PFS) | 2 years
Time to intracranial (IC) progression | 2 years
Median Intracranial Duration of Response (DOR) | 2 years
  The distribution function of DOR will be estimated using the Kaplan-Meier method
Median extra-cranial PFS | 2 years
  Extra-cranial PFS will be defined as the time from the start of study drug treatment to the date of the first documented progression at an extra-cranial site or death. The distribution of PFS will be estimated using the Kaplan-Meier method.
Median Overall Survival | 2 years
Toxicity assessed using CTCAE v4.0 criteria | 2 years
Intracranial Objective Response Rate (ORR) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ibiayi Dagogo-Jack, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts general Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Dagogo-Jack I, Oxnard GR, Evangelist M, Digumarthy SR, Lin JJ, Gainor JF, Murphy JF, Rabin MS, Heist RS, Muzikansky A, Shaw AT. Phase II Study of Lorlatinib in Patients With Anaplastic Lymphoma Kinase-Positive Lung Cancer and CNS-Specific Relapse. JCO Precis Oncol. 2022 May;6:e2100522. doi: 10.1200/PO.21.00522. PMID 35584349